CLINICAL TRIAL: NCT04731896
Title: Early Versus Late Amniotomy During Labor Induction in Women With Bishop's Score of ≥ 6 : a Randomized Trial
Brief Title: Early Versus Late Amniotomy During Labor Induction in Women With Bishop's Score of ≥ 6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ahmed Halouani, MD, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTuniselmanar2
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Labor, Induced; Amniotomy
Keywords: labor; Amniotomy; induction
MeSH Terms: interventions — Amniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late Amniotomy (No Intervention): Initiating induction of labor with oxytocin infusion followed by amniotomy 4-6 hours later
- Early Amniotomy (Active Comparator): Early amniotomy initiating induction of labor followed by oxytocin infusion 30 minutes later
  Interventions: Procedure: Amniotomy

INTERVENTIONS:
Procedure: Amniotomy — artificial rupture of the amniotic sac
  Arms: Early Amniotomy

SUMMARY:
Labor induction is the stimulation of uterine contractions during pregnancy, before labor begins on its own to achieve a vaginal birth.

A health care provider might recommend labor induction for various reasons: primarily when there's concern for a mother's health or a baby's health.

Combined with oxytocin infusion, amniotomy is commonly used in the induction of labor. However the perfect timing of amniotomy is still unknown.

The aim of this study is to determine whether the early amniotomy followed by oxytocin, or initiating induction of labor with oxytocin followed by late amniotomy, is effective to reach active phase of labor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Full term (36 weeks and 3 days of gestation reached)
* Singletion gestation in cephalic presentation
* Bishop score of ≥ 6

Exclusion Criteria:

* Prior uterine surgery, previous cesarean section
* Ruptured membranes
* Spontaneous labor
* Multifetal pregnancy
* Dystocic presentation
* Fetal head not fixed at pelvic brim
* Macrosomia
* Hydramnios
* Severe fetal growth restriction
* Major fetal anomaly
* Women with HIV, hepatitis C, hepatitis B
* Women with medical conditions contraindication to a vaginal delivery
* Women with COVID-19 infection

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time to active phase of labor | At delivery
  Total time from initiation oxytocin infusion to reaching 5 cm cervical dilation

SECONDARY OUTCOMES:
Cesarean delivery rate | At delivery
  Rate of cesarean section
Time to vaginal delivery | At delivery
  Total time from initiation of labor induction to vaginal delivery
Maternal outcomes | From inclusion to discharge, up to 2 weeks
  Intrapartum and postpartum fever, postpartum haemorrhage, chorioamnionitis, endometritis
Fetal and neonatal outcome | From inclusion to discharge, up to 2 weeks
  Fetal distress, birth asphyxia, acidosis, sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Mongi Slim la Marsa, Tunis, La Marsa, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years from 01/01/2022